CLINICAL TRIAL: NCT00005488
Title: Common Variants in Candidate Genes and Premature MI Risk
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5004; R01HL056931 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2005-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Myocardial Infarction
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Myocardial Infarction

SUMMARY:
To examine the impact of an interaction between common genetic susceptibility markers and environmental exposures on risk for early onset myocardial infarction in cases with myocardial infarction and matching controls.

DETAILED DESCRIPTION:
BACKGROUND:

Inherited factors play a role in the pathogenesis of myocardial infarction (MI), and there is growing interest in identifying common genetic susceptibility markers that interact with common environmental exposures to contribute to the occurrence of myocardial infarction (MI) in the population.

DESIGN NARRATIVE:

The study had a case-control design. The preliminary data addressed the contribution of common genetic and environmental factors to the risk of MI among women under 45 years of age. Those data showed that common polymorphisms in genes coding for two clotting factors, coagulation Factor V and coagulation Factor II, were risk factors for MI only among cigarette smokers in this sample. These relationships, and others observed, provided strong evidence of gene-environment interactions between thrombotic and atherosclerotic factors in early-onset MI. One intent was to determine whether the risk of early-onset MI was related to interactions between environmental factors (e.g., cigarette smoking, exercise, alcohol consumption) and common polymorphisms in genes coding for thrombotic factors (coagulation Factor V, coagulation Factor II, plasminogen activator inhibitor-1, and beta-fibrinogen) and atherosclerotic factors (the adhesion molecule E-selectin and metalloproteinase stromelysin-1; the lipid metabolism enzymes paraoxinase, lipoprotein lipase, cholesterol ester transfer protein; and the apolipoproteins apolipoprotein E and apolipoprotein B). Additionally, there were plans to determine whether the risk of early-onset MI was related to interactions between plasma lipoprotein(a) levels (which were largely genetically determined) and environmental risk factors and/or polymorphisms in the candidate genes. Interactions among candidate polymorphisms were also assessed.

Newly-diagnosed cases of MI and controls will be interviewed in person to assess medical and behavioral characteristics related to MI risk. A venous blood sample will be obtained and processed into aliquots of plasma and white cells. DNA extracted from the white cells will be tested using the polymerase chain reaction (PCR), PCR/restriction fragment length polymorphisms (RFLP), and oligonucleotide ligation assays to determine the genotypes of interest. Plasma will be tested for lipid, lipoprotein, and homocysteine concentrations. Analyses will address both the overall association between the genotypes and MI risk, along with posited gene-environment and gene-gene interactions.

ELIGIBILITY:
No eligibility criteria

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1998-07; Study Completion 2002-08

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Schwartz — University of Washington